CLINICAL TRIAL: NCT04003935
Title: Effects of Long-term Consumption of Two Plant-based Dietary Supplements on Low-grade Inflammation, Cardiovascular Disease Prevention and Circulating Micronutrients in a Cohort of Elderly Volunteers
Brief Title: Juice Plus Inflammaging and Cardiovascular Disease Prevention Study
Status: Terminated | Type: Observational
Why Stopped: One of the 2 nutritional products is reformulated and withdrawn from the market
Sponsor: Green Beat (Other)
Collaborators: Medical University of Graz (Other)
Responsible Party: Principal Investigator, Lamprecht Manfred PhD, PhD, Principal Investigator, Green Beat
Other Study IDs: 31-242 ex 18/19
Record Dates: First submitted 2019-06-04; First posted 2019-07-01 (Actual); Last update posted 2020-05-29 (Actual); Status verified 2020-05

CONDITIONS: Overweight or Obesity
Keywords: low-grade inflammation; aging; CVD prevention
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum samples stored for future micronutrient analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Control: Continuing habitual diet and lifestyle.
- Active 1: Ingestion of a macro- and micro-nutrient rich shake, otherwise continuing habitual diet and lifestyle.
  Interventions: Other: Juice Plus+ Complete
- Active 2: Ingestion of an encapsulated vitamin and phytonutrient supplement, otherwise continuing habitual diet and lifestyle.
  Interventions: Dietary Supplement: Juice Plus+ Premium

INTERVENTIONS:
Other: Juice Plus+ Complete — Plant-based smoothie; maintaining habitual diet.
  Groups: Active 1
Dietary Supplement: Juice Plus+ Premium — Fruit and vegetable juice concentrate; maintaining habitual diet.
  Groups: Active 2

SUMMARY:
Low- grade inflammation is a pathological feature of a wide range of chronic conditions, including the metabolic syndrome, cardiovascular diseases (CVD) and the accelerated reduction in bone density. Previous research shows that diets rich in fruits and vegetables can reduce chronic inflammation. To date there is no data on multiyear clinical interventions assessing the effect of plant-based dietary supplements on low-grade inflammation, cardiovascular disease prevention and indicators of biological aging, including individuals' cognitive function. In this study, the investigators are thus exploring whether separate ingestions of two plant-based nutritional products over 2 years, are able to modulate low-grade inflammation, parameters of CVD prevention, circulating micronutrients, upper respiratory tract- and gastro-intestinal symptoms, quality of life, indicators of biological aging, and cognitive function in overweight seniors.

DETAILED DESCRIPTION:
Inflammation is a central component of innate (non-specific) immunity. The termination of inflammation is an active process involving cytokines and anti-inflammatory mediators like lipids and micronutrients. Inflammation acts as both, 'friend and foe'; it is an essential component of immunosurveillance and host defense, but a chronic low-grade inflammatory state is a pathological feature of a wide range of chronic conditions, such as the metabolic syndrome or cardiovascular diseases (CVD). In addition, low-grade inflammation and oxidative stress are often associated with increased body fat mass, obesity but also accelerated reduction in bone density.

There is a substantial amount of evidence to suggest that many foods, nutrients and non-nutrient food components modulate inflammation both acutely and chronically. Nutritional regimens with adequate intake of micronutrients, vegetables, and fruits, low in sugar and saturated fats, like the Mediterranean diet or a vegetarian dietary regimen, can reduce chronic inflammation and oxidative stress.

To date there is no data on multiyear clinical interventions assessing the effect of plant-based dietary supplements on low-grade inflammation, cardiovascular disease prevention and indicators of biological aging, including individuals' cognitive function. In this study, the investigators are thus exploring whether separate ingestions of two plant-based nutritional products over 2 years, are able to modulate biomarkers of low-grade inflammation and CVD prevention, plasma concentrations of micronutrients, upper respiratory tract- and gastro-intestinal symptoms, quality of life, indicators of biological aging, and cognitive function in an overweight/obese cohort of middle-aged, elderly people.

Volunteers expressing interest to take part in the study, will need to attend a screening visit where their eligibility will be assessed. For participants with confirmed eligibility, they will need to attend a baseline visit and consecutive study visits at 6, 12, 18 and 24 months. Markers of low-grade inflammation and CVD, micronutrients status, respiratory tract symptoms, gastrointestinal symptoms and quality of life will be assessed at baseline, 6, 12, 18 and 24 months. Bone quality and telomere length will be assessed at baseline, 12 and 24 months.

Propensity score approach:

Since this is a long-term trial and in order to maximize adherence to the ingestion of the products, volunteers will be allowed to choose their preferred nutritional product. Instead of using randomization, the investigators have chosen a propensity score (PS) approach which helps to reduce bias with regards to random significances. More specifically, for each participant an individual score based on certain parameters, likely to affect the primary outcomes, will be calculated and will be matched with another participant with the same PS across the three groups. PS matching will be implemented without replacement and setting the caliper equal to 0.025. Furthermore, to ensure an adequate number of matching PSs between groups, about a 3-fold number of subjects needed to enter the study, will be pre-screened.

Sample size:

With a sample size of 20 subjects per group (total sample size = 60), the disjunctive power for testing each primary endpoint (i.e., the probability of establishing a significant effect in supplementation-control or between-supplementation comparisons) is 78%, 51%, 97% for TNF-α, homocysteine and vitamin C (1st ranked parameter for each co-primary outcome), respectively.

In addition, it is estimated to have a maximum drop-out rate of 30% over 2 years. In order to ensure balanced distribution of subjects across the three different groups, the investigators will also stratify for gender and age. Based on this sample size calculation and in order to meet the stratification standards, 30 subjects will be recruited to be allocated to each group, corresponding to a total N of 90 subjects.

Statistical analysis:

Statistical analysis will be performed by using SPSS for Windows software, version 22.0. Metric data will be presented as mean ± SD. Statistical significance is set at P < 0.05. The Shapiro-Wilk test will be used to determine normal distribution. To check homogeneity of variances the Levene test will be used. Comparisons of mean values of metric baseline data between the 3 groups will be done by analysis of variance, ANOVA.

If data are normally distributed and variance homogeneity is fulfilled, all metric analytes from blood (low-grade inflammation markers, CVD-prevention markers, micronutrients, telomer length, clinical chemistry etc) will be analyzed by one- and two-factorial (either 'time' or 'time x treatment') repeated measures analysis of variance (ANOVA) and co-variance (ANCOVA, e.g. diet/dietary inflammatory index (DII), exercise), within each group and between groups. Student's t-test for paired samples will be used for within group analysis as soon as 6-month data are available. For post-hoc analyses the Bonferroni(-Holm) correction and/or Tukey´s post-hoc test will be used.

If it is not possible to use metrical data, non-parametric tests will be used like the Friedman Test (within group) and the Kruskal Wallis test (between groups). If differences between groups reach significance the Tukey's post hoc test, the Bonferroni correction or the Bonferroni-Holm-method (for non-parametric data) will be used to determine the localization of the differences.

A comprehensive correlation analyses to compute relations within each outcome-category and between the different outcome-categories will be conducted, also the PS-categories will be included into these correlation analyses.

ELIGIBILITY:
Inclusion Criteria:

* 90 male and female subjects
* age: 50 - 80 years
* post- or peri-menopausal
* Smokers and non-smokers
* BMI 25 to 40 kg/m2
* Dietary Inflammatory Index, DII: 0 to +10
* Fruit and vegetable intake <4 servings/d
* Adherence to a 6-week "wash-out" period
* Since the intervals between blood drawings are long (6 months), a temporary intake (e.g for a few days, one or two weeks) of some excluded drugs and food supplements does not necessarily mean exclusion from the study

Exclusion Criteria:

* Age <50 and >79.9 years
* Dietary Inflammatory Index, DII: - 0.1 to -10
* Subjects with any kind of food allergy or histamine intolerance
* Aversion to stop the intake of nutritional supplements and food, that could interfere with the study outcome
* Food supplements, functional foods and dietetic products with anti-inflammatory or redox-biological relevance like omega-3 fatty acids, plant/herbal extracts/concentrates, vitamin- and mineral supplements
* Fruit and vegetable intake >3 servings per day
* Hypertension, starting with grade 2 according to the classification of the European Society of Hypertension: systolic blood pressure > 160 mmHg, diastolic blood pressure >100 mmHg
* Medication: any anti-inflammatory medication and medication with relevant antioxidant properties, blood pressure lowering medication, psychotropic drugs, immunosuppressives, cytostatics, anticoagulants, contraceptives, diuretics, pain medication
* Clinically relevant infectious disease
* Diabetes mellitus type I and type II
* Auto-immuno diseases
* Any stents and Coronary artery diseases (CAD)
* Cancer patients
* Pregnancy

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Overweight and obese subjects with a higher probability of a low-grade inflammatory status compared to lean people.
Sampling Method: Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-05-27 (Actual); Study Completion 2020-05-27 (Actual)

PRIMARY OUTCOMES:
Concentration changes in biomarkers of low-grade inflammation | 24 months
  TNF-α, TNFsR2, TNFsR1, RANTES/ CCL5, IL-1β, osteoprotegerin (OPG)
Plasma concentration changes in biomarkers of CVD | 24 months
  Homocysteine, oxLDL, Chol, HDL, LDL, Triglycerides, Apo A1, HOMA-IR, Insulin, Glucose, HbA1c, osteocalcin
Efficacy of micronutrients' absorption | 24 months
  Vitamin C, α-carotene, lycopene, ß-cryptoxanthin, α-tocopherol, vitamin A (retinol), ß-carotene, lutein/zeaxanthin, γ-tocopherol, vitamin D, vitamin K1, vitamin K2 (MK-7), matrix gla protein (MGP)

SECONDARY OUTCOMES:
Wisconsin upper respiratory symptoms survey (WURSS) | 24 months
  This is an exploratory questionnaire, consisting of 21 questions and collects information on respiratory tract symptoms.
Gastrointestinal symptoms survey (GISS-14) | 24 months
  This is a questionnaire consisting of 14 questions and is an exploratory assessment of overall gastrointestinal symptoms.
Quality of life | 24 months
  Quality of life will be assessed through the Short Form Survey (SF-36). This is a questionnaire, consisting of 36 questions and 8 scales namely: 1) Physical functioning, 2) Role limitations due to physical health, 3) Role limitations due to emotional problems, 4) Energy/fatigue, 5) Emotional well-being, 6) Social functioning, 7) Pain and 8) General Health.
  All questions are scored on a scale from 0 to 100, with higher scores representing a better health state.
Body mass assessment | 24 months
  Dincl, Dexcl
Anthropometrics | 24 months
  waist circumference, mid arm muscle circumference, BMI, waist/hip ratio

OTHER OUTCOMES:
Cognitive function test | 24 months
  A total CFD-index can be calculated across all domains, taking into account the following dimensions: Expressive language, executive function, verbal long-term memory, attention, and perceptual motoric function
Bone quality | 24 months
  Stiffness index via ultrasound measures
Telomere length | 24 months
  PBMCs, T/S

CONTACTS AND LOCATIONS:
Overall Officials: Manfred Lamprecht, PhD, Principal Investigator — Medical University of Graz
Locations (2):
- Austria (2):
  - Institute of Pathophysiology and Immunology, Graz, Styria
  - Green Beat, Graz

IPD SHARING:
Plan to Share IPD: Undecided